CLINICAL TRIAL: NCT00374088
Title: Attenuation of Myocardial Dysfunction by N-Acetylcysteine in Infants Undergoing Arterial Switch Procedure
Brief Title: N-Acetylcysteine in Neonatal Congenital Heart Surgery (INACT Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Ranjit Aiyagari, Clinical Assistant Professor of Pediatrics, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRBMED No.: 2004-851
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Results first posted 2012-01-19 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2011-12

CONDITIONS: Transposition of Great Vessels; Congenital Heart Disease
Keywords: N-acetylcysteine; Myocardial dysfunction; Transposition of the Great Arteries
MeSH Terms: conditions — Transposition of Great Vessels; Heart Defects, Congenital | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): These patients receive a placebo infusion of D5W prior to and after surgery
  Interventions: Drug: Placebo
- N-Acetylcysteine (Experimental): These patients receive a loading dose of N-Acetylcysteine 100 mg/kg in D5W IV 1 hour prior to surgery. They receive a maintenance infusion of N-Acetylcysteine 10 mg/kg/hr in D5W IV for 24 hours after surgery.
  Interventions: Drug: N-acetylcysteine

INTERVENTIONS:
Drug: N-acetylcysteine — Loading dose: Subjects randomized to IV NAC will receive a total loading dose of 100 mg/kg of 10% (100 mg/mL) solution. Acetadote is supplied as a 20% solution (200 mg/mL) and will be diluted 1:1 with an equal volume of D5W. The volume of the loading dose will be 1 mL/kg, anticipated to be 2.5-5 mL in our patient population. The loading dose will be administered over 1 hr beginning 1 hr prior to the patient's OR time. Subjects in the placebo group will receive 1 mL/kg of D5W over 1 hr.
  Maintenance infusion: Subjects randomized to IV NAC will receive an infusion of 10 mg/kg/hr of 10% (100 mg/mL) solution for 24 hrs, starting in the OR after weaning from CPB. Acetadote is supplied as a 20% solution (200 mg/mL) and will be diluted 1:1 with an equal volume of D5W. The volume of the maintenance infusion will be 0.1 mL/kg/hr, anticipated to be 0.25-0.5 mL/hr in our patient population. Subjects in the placebo group will receive 0.1 mL/kg/hr of D5W for 24 hrs.
  Arms: N-Acetylcysteine
Drug: Placebo — D5W bolus prior to surgery and D5W infusion after surgery in an equal volume to the drug arm.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether intravenous N-acetylcysteine (also known as Acetadote), an antioxidant medication that has been used for years to treat Tylenol overdose, helps prevent heart dysfunction in the early postoperative period following congenital heart surgery. Children undergoing major heart surgery, such as the arterial switch operation, routinely develop temporary heart dysfunction in the first 12-24 hours after surgery. This heart dysfunction may be severe and contributes to an increased risk for death or prolonged hospitalization. Current standard treatments include intravenous medications such as dopamine, epinephrine, and vasopressin that support your child's blood pressure and heart function. Unfortunately, high doses of these medications have the potential to cause severe side effects including loss of fingers and toes, liver and kidney dysfunction, and heart rhythm abnormalities. Our goal is to find a way to reduce heart dysfunction after major heart surgery in order to promote a smoother postoperative period, and reduce the risks associated with heart operations in children.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, blinded study of intravenous N-acetylcysteine (NAC) for the prevention of postoperative myocardial dysfunction and apoptosis in infants undergoing arterial switch for D-transposition of the great arteries. Subjects will be age 0-3 months, and no distinctions will be made based on gender or race. Infants operated before 36 weeks post-conceptional age or with birth weight less than 1.8 kilograms will be excluded. Informed consent will be obtained from the patient's parent by one of the investigators in the hospital before the infants undergo surgery.

Subjects will be randomized based on a block randomization scheme to receive placebo or NAC infusion, starting with a loading dose 1 hour prior to surgery. If there is any concern by the ICU physician that the patient is developing toxicity to the medicine, the study drug will be discontinued and the patient removed from the study. Patients will have a thermodilution catheter placed during surgery for postoperative direct measurement of cardiac output. Endomyocardial biopsy will be performed by the surgeon pre- and post-bypass for measurement of markers of apoptosis. Postoperatively, patients will continue to receive an infusion of IV NAC for 24 hours. Blood draws will be through existing arterial and central venous catheters. Serum labs collected will include serial lactate values (already collected routinely), liver and renal function tests, CK-MB and troponin-I levels as a marker of myocardial injury, and S100b level as a marker of brain injury. Total additional blood removed for research purposes will be less than 15 mL. Cardiac output will be measured serially by thermodilution. Serial transthoracic echocardiography will be used to determine left ventricular function. Inotropic score, duration of mechanical ventilation, length of ICU stay, and length of hospitalization will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* All patients transferred to or born at C.S. Mott Children's Hospital between 0 and 3-months-old undergoing ASO for d-TGA or anatomic variants (including double-outlet right ventricle with transposition physiology).

Exclusion Criteria:

* Less than 36-weeks post-conceptional age at the time of enrollment
* Birth weight less than 1800 grams;
* Evidence of significant renal, hepatic, or neurological dysfunction
* Additional significant cardiac lesions other than patent ductus arteriosus, isolated ventricular septal defect, simple coarctation, and/or atrial septal defect
* Preoperative extracorporeal membrane oxygenation (ECMO).

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2005-02; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ranjit M Aiyagari, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Wernovsky G, Wypij D, Jonas RA, Mayer JE Jr, Hanley FL, Hickey PR, Walsh AZ, Chang AC, Castaneda AR, Newburger JW, Wessel DL. Postoperative course and hemodynamic profile after the arterial switch operation in neonates and infants. A comparison of low-flow cardiopulmonary bypass and circulatory arrest. Circulation. 1995 Oct 15;92(8):2226-35. doi: 10.1161/01.cir.92.8.2226. PMID 7554206
- [Background] Tossios P, Bloch W, Huebner A, Raji MR, Dodos F, Klass O, Suedkamp M, Kasper SM, Hellmich M, Mehlhorn U. N-acetylcysteine prevents reactive oxygen species-mediated myocardial stress in patients undergoing cardiac surgery: results of a randomized, double-blind, placebo-controlled clinical trial. J Thorac Cardiovasc Surg. 2003 Nov;126(5):1513-20. doi: 10.1016/s0022-5223(03)00968-1. PMID 14666027
- [Background] Braunwald E, Kloner RA. Myocardial reperfusion: a double-edged sword? J Clin Invest. 1985 Nov;76(5):1713-9. doi: 10.1172/JCI112160. No abstract available. PMID 4056048
- [Background] Kofsky E, Julia P, Buckberg GD, Young H, Tixier D. Studies of myocardial protection in the immature heart. V. Safety of prolonged aortic clamping with hypocalcemic glutamate/aspartate blood cardioplegia. J Thorac Cardiovasc Surg. 1991 Jan;101(1):33-43. PMID 1986168
- [Background] Julia P, Kofsky ER, Buckberg GD, Young HH, Bugyi HI. Studies of myocardial protection in the immature heart. III. Models of ischemic and hypoxic/ischemic injury in the immature puppy heart. J Thorac Cardiovasc Surg. 1991 Jan;101(1):14-22. PMID 1986156
- [Background] Itoi T, Lopaschuk GD. Calcium improves mechanical function and carbohydrate metabolism following ischemia in isolated Bi-ventricular working hearts from immature rabbits. J Mol Cell Cardiol. 1996 Jul;28(7):1501-14. doi: 10.1006/jmcc.1996.0140. PMID 8841937
- [Background] Matherne GP, Berr SS, Headrick JP. Integration of vascular, contractile and metabolic responses to hypoxia: effects of maturation and adenosine. Am J Physiol. 1996 Apr;270(4 Pt 2):R895-905. doi: 10.1152/ajpregu.1996.270.4.R895. PMID 8967420
- [Background] Carr LJ, VanderWerf QM, Anderson SE, Kost GJ. Age-related response of rabbit heart to normothermic ischemia: a 31P-MRS study. Am J Physiol. 1992 Feb;262(2 Pt 2):H391-8. doi: 10.1152/ajpheart.1992.262.2.H391. PMID 1539698
- [Background] Young JN, Choy IO, Silva NK, Obayashi DY, Barkan HE. Antegrade cold blood cardioplegia is not demonstrably advantageous over cold crystalloid cardioplegia in surgery for congenital heart disease. J Thorac Cardiovasc Surg. 1997 Dec;114(6):1002-8; discussion 1008-9. doi: 10.1016/S0022-5223(97)70014-X. PMID 9434695
- [Background] Najm HK, Wallen WJ, Belanger MP, Williams WG, Coles JG, Van Arsdell GS, Black MD, Boutin C, Wittnich C. Does the degree of cyanosis affect myocardial adenosine triphosphate levels and function in children undergoing surgical procedures for congenital heart disease? J Thorac Cardiovasc Surg. 2000 Mar;119(3):515-24. doi: 10.1016/s0022-5223(00)70131-0. PMID 10694612
- [Background] Nagashima M, Nollert G, Stock U, Sperling J, Hatsuoka S, Shum-Tim D, Takeuchi K, Nedder A, Mayer JE Jr. Cardiac performance after deep hypothermic circulatory arrest in chronically cyanotic neonatal lambs. J Thorac Cardiovasc Surg. 2000 Aug;120(2):238-46. doi: 10.1067/mtc.2000.106984. PMID 10917937
- [Background] Ahola T, Fellman V, Laaksonen R, Laitila J, Lapatto R, Neuvonen PJ, Raivio KO. Pharmacokinetics of intravenous N-acetylcysteine in pre-term new-born infants. Eur J Clin Pharmacol. 1999 Nov;55(9):645-50. doi: 10.1007/s002280050687. PMID 10638393
- [Background] Perry HE, Shannon MW. Efficacy of oral versus intravenous N-acetylcysteine in acetaminophen overdose: results of an open-label, clinical trial. J Pediatr. 1998 Jan;132(1):149-52. doi: 10.1016/s0022-3476(98)70501-3. PMID 9470017
- [Background] Andersen LW, Thiis J, Kharazmi A, Rygg I. The role of N-acetylcystein administration on the oxidative response of neutrophils during cardiopulmonary bypass. Perfusion. 1995;10(1):21-6. doi: 10.1177/026765919501000105. PMID 7795309
- [Background] Arstall MA, Yang J, Stafford I, Betts WH, Horowitz JD. N-acetylcysteine in combination with nitroglycerin and streptokinase for the treatment of evolving acute myocardial infarction. Safety and biochemical effects. Circulation. 1995 Nov 15;92(10):2855-62. doi: 10.1161/01.cir.92.10.2855. PMID 7586252

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients not treated with N-acetylcysteine
- N-acetylcysteine: Patients treated with N-acetylcysteine
Period: Overall Study
Arm/Group | Placebo | N-acetylcysteine
Started | 10 | 11
Completed | 9 | 10
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | N-acetylcysteine | Total
Number analyzed (Participants) | 10 | 11 | 21
Age Continuous [Mean (Standard Deviation); unit: years] | 0.02 (0.007) | 0.02 (0.006) | 0.02 (0.007)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 5 | 8 | 13
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Maximum Decline in Measured Cardiac Output
Description: Serial cardiac output was measured by thermodilution. The outcome of maximum decline in indexed cardiac output from 1 hour postoperative to lowest output within 24 hours postoperative was then calculated and compared between NAC and placebo groups.
Time Frame: 24 hours
Population: Patients in which the surgeon was technically able to place a 4 French thermodilution catheter into the pulmonary artery at the time of surgery had cardiac output measured.
Measure: Mean (Standard Deviation); unit: L/min/m2
Arm/Group | Placebo | N-acetylcysteine
Number analyzed (Participants) | 9 | 10
L/min/m2 | 0.68 (0.59) | 0.29 (0.56)

2. Post Hoc Outcome: Max Creatinine
Description: Maximum serum creatinine over first 3 days postoperative.
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | N-acetylcysteine
Number analyzed (Participants) | 9 | 10
mg/dL | 0.99 (0.44) | 0.74 (0.24)

3. Post Hoc Outcome: Urine Output
Description: Total urine output over the first 24 hours postoperative
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | N-acetylcysteine
Number analyzed (Participants) | 9 | 10
mL | 96 (54) | 176 (55)

ADVERSE EVENTS:
Time Frame: Duration of hospitalization
Description: Duration of hospitalization varied by patient
Arm/Group | Placebo | N-acetylcysteine
Serious Adverse Events (participants affected / at risk) | 1/10 | 2/11
Other Adverse Events (participants affected / at risk) | 4/10 | 7/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | N-acetylcysteine (N=11)
Bleeding requiring surgical re-exploration (Surgical and medical procedures) | 0 (0) | 1 (1) — Patient underwent an arterial switch operation. Postoperative course had been marked by significant coagulopathy and mediastinal bleeding. Mediastinal exploration for probable cardiac tamponade. (N-acetylcysteine arm)
Grade II bleeds on head ultrasound (Cardiac disorders) | 1 (1) | 0 (0) — Crainial ultrasound performed secondary to his hemodynamic instability. Demonstrated bilateral grade 2 intraventricular hemorrhage. Cardiac surgery delayed. At discharge neurological exam remains normal without any focal neurological symptoms,
Patient placed on ECMO in operating room (Surgical and medical procedures) | 0 (0) | 1 (1) — Patient placed on ECMO in operating room after inability to wean from cardiopulmonary bypass, following surgical kinking of left coronary artery and multiple revisions of anastomosis. Patient successfully decannulated from ECMO 4 days later.
OTHER ADVERSE EVENTS (reported when occurring in more than 2.3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | N-acetylcysteine (N=11)
Junctional Ectopic Tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Persistent fevers (Infections and infestations) | 0 (0) | 1 (1) — Positive cultures requiring 10 day antibacterial therapy
Hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0) — Low glucose, treated and patient recovered the following day.
Poor urine output (Renal and urinary disorders) | 1 (1) | 0 (0) — Dialysis required for 5 days. Patient recovered.
Venous congestion of left leg (Vascular disorders) | 1 (1) | 0 (0)
SVT (Cardiac disorders) | 1 (1) | 2 (2)
Seizures (Nervous system disorders) | 0 (0) | 1 (1)
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes